CLINICAL TRIAL: NCT00679536
Title: Allogeneic Transplantation for Pediatric Leukemias With Unrelated Donors Using Fludarabine, Busulfan, 400 cGy Total Body Irradiation, and Thymoglobulin
Brief Title: Allogeneic Transplantation for Pediatric Leukemias With Unrelated Donors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Sonali Chaudhury, MD, PI, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT 0208
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Leukemia
Keywords: Reduced Toxicity; Toxicity; Event Free Survival; Graft vs Host Disease
MeSH Terms: conditions — Leukemia; Graft vs Host Disease | interventions — Busulfan; fludarabine; fludarabine phosphate; thymoglobulin; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All patients on this trial will receive a conditioning regimen of Busulfan, Fludarabine, Anti-Thymocyte Globulin and Total Body Irradiation (400 cGy)
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Thymoglobulin; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: Busulfan — Patient will receive a Test Dose of Busulfan on either Day -10 or Day -9. Patient will receive their Regimen Dose of Busulfan on Day -5 to Day -2. The regimen dose of Busulfan will be based off of the findings from their Test Dose.
  Other Names: IV Busulfex
Drug: Fludarabine — Patient will receive Fludarabine from Day -6 to Day -2. The dose of Fludarabine will be 30 mg/m^2/day.
  Other Names: Fludara
Drug: Thymoglobulin — The patient will also receive Thymoglobulin (rabbitATG) on Day -4 to Day -2. Each dose of rabbitATG will be 1.5 mg/kg/day.
Radiation: Total Body Irradiation — On Day -1 the patient will receive a total of 400 cGy of Total Body Irradiation.

SUMMARY:
The study proposes the use of Fludarabine, Busulfan, Anti Thymocyte Globulin Rabbit (ATG) and Total Body Irradiation as a preparative regimen before hematopoietic stem cell transplant from unrelated donor peripheral blood stem cells (PBSC). The hypothesis states that the 100 day mortality after this type of transplant will be significantly below the accepted standards, which is about 30% for unrelated donors.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the toxicity (as measured as 100 day survival) after hematopoietic stem cell transplant from an unrelated donor with a novel preparative regimen of Fludarabine, Busulfan, Anti-Thymocyte Globulin, and Total Body Irradiation for pediatric patients with leukemia. The secondary objectives are to evaluate the relapse-free and overall survival after hematopoietic stem cell transplant as well as to evaluate the incidence of acute and chronic graft-versus-host disease after this preparative regimen.

ELIGIBILITY:
Inclusion Criteria:

* Ages 0-21
* AML in one of the following stages:

  * Having preceding myelodysplasia (MDS)
  * High Risk cytogenetics
  * Requiring > 2 cycles chemotherapy to obtain complete remission
  * High allelic ratio FLT3/ITD+,
  * Standard risk cytogenetics with positive MRD at end of Induction
  * Second or greater CR
  * First relapse with < 25% blasts in bone marrow
  * With therapy-related AML whose prior malignancy has been in remission for at least 12 months
* ALL in one of the following stages:
* High risk first remission, defined as:

  * Ph+ ALL; or,
  * MLL rearrangement with slow early response [defined as having M2 (5-25% blasts) or M3 (>25% blasts on bone marrow examination on Day 14 of induction therapy)]; or,
  * Hypodiploidy (< 44 chromosomes or DNA index < 0.81); or,
  * End of induction M3 bone marrow; or,
  * End of induction M2 marrow or MRD>1% with M2-3 marrow or MRD>1% at Day 42.
  * High-risk infant ALL defined as age <6 months at diagnosis with MLL (11q23) translocation.
* High risk second remission, defined as:

  * Bone marrow relapse < 36 months from induction; or >36 mths if a matched sibling donor is available
  * T-lineage relapse at any time; or,
  * Very early isolated CNS relapse (<18 months from diagnosis); or,
  * Slow reinduction (M2-3 at Day 28) after relapse at any time.
* Any third or subsequent CR.
* Biphenotypic or undifferentiated leukemia in any CR or if in first relapse must have < 25% blasts in bone marrow
* MDS at any stage; prior therapies allowed
* CML in chronic or accelerated phase; prior therapies allowed
* Patient also must have the following organ requirements:

  * Adequate renal function defined as serum creatinine <2x normal, or creatinine clearance > 40 ml/min/m^2 or 70 ml/min.
  * Adequate liver function as defined by total bilirubin less than or equal to 2 times normal and AST and ALT less than or equal to 4 times normal.
  * Adequate cardiac function as defined by: shortening fraction > 24% by echocardiogram, or ejection fraction > 30% by radionuclide angiogram.
  * Adequate pulmonary function as defined by DLCO, FEV1/FVC > 60% by pulmonary function tests. For children who are uncooperative for PFTs and have no evidence of dyspnea at rest or exercise intolerance, pulse oximetry > 94% on room air is considered acceptable, with a normal chest xray.
  * Adequate venous access; a double lumen central vascular access device or its equivalent and an additional PICC line will be required for all patients.
* Women of childbearing potential and sexually active males should use effective contraception while on study.

Exclusion Criteria:

* Inability to give informed consent or assent
* Inability to obtain a suitable donor
* Patient who is HIV-positive
* Patient who has active Hepatitis B
* Patient who is pregnant
* Patient who is otherwise considered unsuitable for transplant at the discretion of the principal investigator.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the toxicity (as measures by 100 day survival) after hematopoietic stem cell transplant from an unrelated donor with a novel preparative regimen. | 100 day mortality

SECONDARY OUTCOMES:
To evaluate the relapse-free and overall survival after hematopoietic stem cell transplant with Fludarabine/Busulfan/ATG/TBI preparative regimen for pediatric patients with leukemia. | 5 years
To evaluate the incidence of acute and chronic graft-versus-host disease after hematopoietic stem cell transplant | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Chaudhury, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States